CLINICAL TRIAL: NCT00850265
Title: Rol of Spacer in the Combined Treatment With Extrafine Beclomethasone-Formoterol in Stable Asthma
Brief Title: Effect of Spacer in Extrafine Formoterol-Beclomethasone Treatment to Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Requena (Other)
Responsible Party: Miguel Angel Martínez García, Hospital General de Requena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FORM-DPB-extrafine
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Beclomethasone; Extrafine formulation; Spacer; Moderate; Severe; Stable
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spacer (Experimental): Extrafine formoterol plus beclomethasone with spacer
  Interventions: Device: Volumatic spacer
- No Spacer (No Intervention): Extrafine formoterol plus beclomethasone without spacer

INTERVENTIONS:
Device: Volumatic spacer — A spacer is a plastic device to inhaler medication
  Arms: Spacer

SUMMARY:
Combined inhaled treatment with long acting adrenergics and steroids in an unique inhaler plays an important role in the management of non-mild asthma. Some studies have demonstrated that the use of spacers achieve better lung deposition and decrease the number of side effects. Recently a new combined treatment for asthma has been developed (extrafine formoterol plus beclomethasone dipropionate). The small size of the extrafine particles of this new combination get the small airway and theorically improve their positive effect. Some authors have stated that the use of a spacer with extrafine particle could decrease the effectiveness of this treatment due to the adhesion of particles on the walls of the spacer because of the electrostatic characteristics of plastic spacers. However, there are no clinical or functional studies demonstrating the role of this phenomena in the control of asthmatic patients. The investigators' hypothesis is that the benefit of using spacers with this new treatment is at least equal in magnitude than the loss of efficacy because of the adhesion of particles on the wall of the spacer and then the investigators hypothesized that the use of spacer with extrafine formoterol-beclomethasone do not suppose a decrease in clinical or functional control in stable moderate-severe asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe asthma
* Stable asthma
* 18-75 years old

Exclusion Criteria:

* Exacerbation of asthma
* Instability with the study treatment
* Other cardiopulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | at 3 months

SECONDARY OUTCOMES:
Peak Flow | at 3 months
Asthmatics Symptoms | at 3 months
Side effects | at 3 months
Inhalation technique | at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Requena, Requena-Valencia, Valencia, Spain